CLINICAL TRIAL: NCT00626288
Title: A Randomised Controlled Multicenter Trial Assessing the Efficacy and Safety of Mesalazine Therapy in Patients With Irritable Bowel Syndrome.
Brief Title: Mesalazine Therapy in Patients With Irritable Bowel Syndrome
Acronym: IBS-02/07
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IBS
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: Mesalazine in Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Mesalazine cpr 800 mg t.i.d. for 12 weeks
  Interventions: Drug: Mesalazine
- B (Placebo Comparator): Placebo cpr t.i.d. for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesalazine — Mesalazine 800mg t.i.d. 12 weeks
  Other Names: Pentacol 800, Sofar
  Arms: A
Drug: Placebo — Placebo cpr, t.i.d. 12 weeks
  Arms: B

SUMMARY:
The purpose of this study is to determine whether Mesalazine is effective in the treatment of the abdominal discomfort or pain of Irritable Bowel Syndrome patients.

DETAILED DESCRIPTION:
The present study is a prospective, double blind, randomised, multicenter trial designed to study the efficacy of mesalazine treatment on symptoms of IBS. In a subgroup of patients the efficacy of this treatment will be also assessed on low-grade inflammation. We expect to confirm that mesalazine treatment reduces the number and activation of inflammatory cells in the colonic mucosa of IBS patients, thus providing the rationale for the assessment of this treatment on symptoms of IBS.

ELIGIBILITY:
Inclusion Criteria:

* IBS patients with positive diagnosis inclosing Rome III criteria

Exclusion Criteria:

* Any organic or metabolic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2007-12; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
"Responder" is the patient who affirmatively answers on at least 50% of the weekly question:"Did you have satisfactory relief of your abdominal discomfort or pain during the last week?". | 3 months

SECONDARY OUTCOMES:
"Responder" is the patient who affirmatively answers on at least 50% of the weekly question:"Did you have satisfactory relief of your overall IBS symptoms during the last week?". VAS scale IBS-QoL questionnaire and SF-36 questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Corinaldesi, Professor, Study Director — Azienda Ospedaliero-Universitaria di Bologna Policlinico S.Orsola Malpighi; Barbara Giovanni, Doctor, Principal Investigator — Azienda Ospedaliero-Universitaria di Bologna Policlinico S.Orsola Malpighi
Locations (22):
- Italy (22):
  - Ospedali Riuniti Torrette, Ancona, Ancona
  - Azienda Ospedaliero-Universitaria S.Orsola Malpighi, Bologna, Bologna
  - U.O. Medicina Interna- Osp. S.S.Annunziata, Cento, Ferrara
  - Azienda Sanitaria Unità Locale di Ferrara- Ospedale del Delta, Lagosanto, Ferrara
  - Opera Padre Pio, Foggia, Foggia
  - Azienda Ospedaliera Polo Universitario L.Sacco, Milan, Milano
  - Policlinico S.Donato, San Donato, Milano
  - A.O.U. Policlinico Seconda Università, Napoli, Napoli
  - Policlinico, Napoli, Napoli
  - U.O. Gastroenterologia Universitaria, Pisa, Pisa
  - Ospedale S. Maria delle Croci, Ravenna, Ravenna
  - Azienda Ospedaliera San Camillo-Forlanini, Roma, Roma
  - Ospedale Universitario Sant'Andrea, Roma, Roma
  - Università Campus Biomedico, Roma, Roma
  - Ospedale S. Andrea, Vercelli, VC
  - Ospedale Umberto I Venezia-Mestre, Mestre, Venezia
  - Policlinico G.B. Rossi, Verona, Verona
  - Azienda ULSS 1, Belluno
  - Azienda Ospedaliero-Universitaria S. Orsola Malpighi, Bologna
  - Ospedale SS. Annunziata, Chieti
  - Ospedale Careggi, Florence
  - Fondazione IRCCS Policlinico, Milan

REFERENCES:
- [Background] Barbara G, Wang B, Stanghellini V, de Giorgio R, Cremon C, Di Nardo G, Trevisani M, Campi B, Geppetti P, Tonini M, Bunnett NW, Grundy D, Corinaldesi R. Mast cell-dependent excitation of visceral-nociceptive sensory neurons in irritable bowel syndrome. Gastroenterology. 2007 Jan;132(1):26-37. doi: 10.1053/j.gastro.2006.11.039. PMID 17241857
- [Background] Barbara G, De Giorgio R, Stanghellini V, Cremon C, Salvioli B, Corinaldesi R. New pathophysiological mechanisms in irritable bowel syndrome. Aliment Pharmacol Ther. 2004 Jul;20 Suppl 2:1-9. doi: 10.1111/j.1365-2036.2004.02036.x. PMID 15335408
- [Background] Barbara G, Stanghellini V, De Giorgio R, Cremon C, Cottrell GS, Santini D, Pasquinelli G, Morselli-Labate AM, Grady EF, Bunnett NW, Collins SM, Corinaldesi R. Activated mast cells in proximity to colonic nerves correlate with abdominal pain in irritable bowel syndrome. Gastroenterology. 2004 Mar;126(3):693-702. doi: 10.1053/j.gastro.2003.11.055. PMID 14988823
- [Background] Barbara G, De Giorgio R, Stanghellini V, Cremon C, Corinaldesi R. A role for inflammation in irritable bowel syndrome? Gut. 2002 Jul;51 Suppl 1(Suppl 1):i41-4. doi: 10.1136/gut.51.suppl_1.i41. PMID 12077063
- [Derived] Barbara G, Cremon C, Annese V, Basilisco G, Bazzoli F, Bellini M, Benedetti A, Benini L, Bossa F, Buldrini P, Cicala M, Cuomo R, Germana B, Molteni P, Neri M, Rodi M, Saggioro A, Scribano ML, Vecchi M, Zoli G, Corinaldesi R, Stanghellini V. Randomised controlled trial of mesalazine in IBS. Gut. 2016 Jan;65(1):82-90. doi: 10.1136/gutjnl-2014-308188. Epub 2014 Dec 22. PMID 25533646